CLINICAL TRIAL: NCT02472431
Title: Effectiveness and Safety of Intracavernosal Administration of Autologous Adipose-Derived Regenerative Cells for Treatment of Erectile Dysfunction
Brief Title: Effectiveness and Safety of Adipose-Derived Regenerative Cells for Treatment of Erectile Dysfunction
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Central Clinical Hospital w/Outpatient Health Center of Business Administration for the President of Russian Federation (Other Government)
Collaborators: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RU-CCH-01-01-15
Record Dates: First submitted 2015-06-09; First posted 2015-06-15 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-11

CONDITIONS: Erectile Dysfunction; Impotence, Vasculogenic
Keywords: ADRC; Adipose-Derived Regenerative Cells; Fat Tissue; Stem Cells; Erectile Dysfunction; Arteriogenic Impotence; Venogenic Impotence; Vasculogenic Impotence; Male Impotence; Male Sexual Impotence
MeSH Terms: conditions — Erectile Dysfunction; Impotence, Vasculogenic | interventions — Lipectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ADRC injection (Experimental)
  Interventions: Other: Intracavernosal administration of autologous ADRC; Procedure: Liposuction; Device: ADRC isolation

INTERVENTIONS:
Other: Intracavernosal administration of autologous ADRC — Subjects will undergo liposuction under local anesthesia. Lipoaspirate will be processed to isolate and concentrate adipose-derived regenerative cells (ADRC). After isolation autologous ADRC suspension will be injected intracavernosally.
Procedure: Liposuction
Device: ADRC isolation — ADRC isolation performed using Celution 800/CRS System (Cytori Therapeutics Inc) according to manufacturer's protocol

SUMMARY:
Autologous adipose-derived regenerative cells (ADRC) extracted using Celution 800/CRS System (Cytori Therapeutics Inc) from a portion of the fat harvested from the patient's front abdominal wall. ADRC will be administered one-time intracavernosally. This is a single arm study with no control. All patients receive cell therapy.

DETAILED DESCRIPTION:
Fat tissue obtainment:

Subjects will undergo liposuction under local anesthesia. In this procedure, Ringer's solution with the anesthetic lidocaine and vasoconstrictor adrenaline infused into the adipose compartment to minimize blood loss and contamination of the tissue by peripheral blood cells. 15 minutes later a hollow blunt-tipped 3 mm cannula introduced into the subcutaneous space through small (0.5 cm) incision. The cannula attached to syringe and under gentle suction moved through the adipose compartment, mechanically disrupting the fat tissue. Aspirate volume - approximately 150-200 cc. Procedure time - 30 minutes.

ADRC isolation:

Aspirated fat tissue placed into sterile vessel which inserted into Celution 800/CRS System (Cytori Therapeutics Inc) - closed system for automated and standardized extraction and concentration of ADRC. Celution 800/CRS System drains excess of fluid from fat tissue and estimate it's volume After that lipoaspirate washed extensively with equal volumes of Ringer's solution to remove blood. At the end of this process System indicates required volume of enzyme reagent (Celase®) which should be added immediately by operator. After enzyme treatment Celution 800/CRS System automatically transfers isolated ADRC into washing compartment where ADRC washed and concentrated in 5 mL suspension. Tissue processing time - approximately 60 minutes. ADRC suspension match all requirements listed in technical documentation for Celution 800/CRS System. Obtained ADRC divided into 2 portions. First portion (0.2-0.5 mL) used for counting, viability and sterility assessment. Second portion placed into sterile insulin syringes with needle size 30 G for injection.

Intracavernosal injection of ADRC:

Tourniquet applied immediately prior to injection at the base of the penis. Penis and surrounding skin treated with antiseptic solution. The injection performed on lateral surface of penis bilaterally proximally into the middle and distal parts of corpus cavernosum. Needle is inserted into the corpus cavernosum at the depth of 5-7 mm. Up to 1.0 ml of ADRC suspension injected per single injection. Equal portions of ADRC suspension injected into both corpora cavernosa. Tourniquet removed 20 minutes after ADRC injection.

ELIGIBILITY:
Inclusion Criteria:

* Patient suffers from erectile dysfunction
* IIEF-5 score less than 21
* Endothelial dysfunction confirmed by EndoPAT measurements
* Patient is familiar with Participant information sheet
* Patient signed informed consent form

Non-inclusion Criteria:

* Contraindications to the local anesthesia or medical history of allergic reactions to local anesthetics
* Patient prescribed for systemic corticosteroids, immunosuppressive drugs, nonsteroidal antiinflammatory drugs, phosphodiesterase-5 inhibitors
* Medical history of penile prosthesis implantation
* Peyronie's disease
* Subcompensated or decompensated forms of chronic diseases of internal organs
* Clinically significant abnormalities in results of laboratory tests
* Any conditions limiting compliance (dementia, neuropsychiatric disease, drug and alcohol abuse etc.)
* Participation in other clinical trials (or administration of investigational drugs) during 3 months prior inclusion
* Patients with malignant tumors including postoperative period, patients receiving chemotherapy and/or radiotherapy.
* Patient's activated partial thromboplastin time exceeds normal levels more than 1,8 times
* Patients prescribed for anticoagulants treatment or patient received anticoagulants at least one hour prior liposuction
* Medical history of heterotopic ossifications
* Patients prescribed for glycoprotein inhibitors treatment
* Patients with infections or septic condition

Exclusion Criteria:

* Patient's refusal from the further participation in trial
* Chronic kidney disease IV- V stages (creatinine clearance < 30 mL/min estimated by Cockcroft-Gault formula)
* Confirmed syphilis, HIV, hepatitis B or C infections
* Patients with hypogonadism

Dropout Criteria:

* Direct indications on immediate initiation of treatment with drugs that have proven effect on erectile function

Ages: 20 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-04; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
SAEs monitoring | 2 weeks after treatment
  Types, probability and severity of treatment emergent serious adverse events (SAEs)
SARs monitoring | 2 weeks after treatment
  Types, probability and severity of treatment emergent serious adverse reactions (SARs)

SECONDARY OUTCOMES:
Quality of life monitoring | Follow up to completion (up to 24 weeks after treatment)
  Quality of life estimated by validated questionnaires: the Short Form (36) Health Survey (SF-36), International Index of Erectile Function (IIEF-5), Sexual Encounter Profile (SEP), Erection Hardness Score (EHS), Global Assessment Question (GAQ)
Penile colour Doppler ultrasonography combined with prostaglandin-E1 injection | Follow up to completion (up to 24 weeks after treatment)
  Colour penile Doppler ultrasonography with intracavernosal injection of prostaglandin-E1 10 ug. Arterial diameter, peak systolic flow velocity, end diastolic flow velocity and resistance index measured before and 15 min after prostaglandin-E1 10ug intracavernosal injection.
Endothelial function assessment | Follow up to completion (up to 24 weeks after treatment)
  Endothelial function assessed by EndoPAT or similar device measurements.
Arterial stiffness assessment | Follow up to completion (up to 24 weeks after treatment)
  Arterial stiffness assessed by EndoPAT or similar device measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Andrey A Pulin, MD, PhD, Principal Investigator — Federal State Budgetary Institution "Central Clinical Hospital with Outpatient Health Center" of the Business Administration for the President of the Russian Federation; Mikhail E Chalyy, MD, PhD, Prof, Principal Investigator — I.M. Sechenov First Moscow State Medical University
Locations (2):
- Russia (2):
  - I.M. Sechenov First Moscow State Medical University, Moscow
  - Federal State Budgetary Institution "Central Clinical Hospital with Outpatient Health Center" of the Business Administration for the President of the Russian Federation; Center for Biomedical Technologies, Moscow